CLINICAL TRIAL: NCT02551341
Title: Randomized Study To Study the Effect of Lung Protective Ventilation (PEEP) Compared With Normal Ventilation (ZEEP) on Lung Function, Kidney Treatment of Sodium and Water, Vasoactive Hormones, Biomarkers of Nephrotoxicity and Haemodynamics in Patients Undergoing Robot-assisted Radical Prostatectomy
Brief Title: Lung Protective Ventilation During Robotic Assisted Prostatectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jørgen Bjerggaard Jensen (Other)
Collaborators: Hospitalsenheden Vest (Other)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEEP-1
Record Dates: First submitted 2015-09-13; First posted 2015-09-16 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Prostate Cancer
Keywords: prostatectomy; robotic
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): normal ventilation
- intervention (Experimental): higher PEEP ventilation
  Interventions: Procedure: higher PEEP ventilation

INTERVENTIONS:
Procedure: higher PEEP ventilation
  Arms: intervention

SUMMARY:
Randomized study investigating the effects of lung protective ventilation (PEEP), as compared with normal ventilation (ZEEP) on lung function, treatment of the renal sodium and water, vasoactive hormones, biomarkers of nephrotoxicity, and the circulation of patients undergoing assisted robotic radical prostatectomy

DETAILED DESCRIPTION:
Protocol Summary

Purpose:

The project will investigate whether a suspected lung protective ventilator therapy in connection with surgery for cancer of the prostate (prostate) have a relevant beneficial effects on lung function, renal function and circulation associated with keyhole surgery performed with surgical robot.

Trial method:

The trial is a randomized study (randomized controlled trials), which are drawn between normal and a suspected lung protective ventilator treatment in connection with the surgical removal of the prostate due to Cancers. Before the operation, collected urine and blood samples and that a study of lung function and circulation as a starting point. During the operation, and in the following two days collected urine and blood samples. Prepare Furthermore, new studies of lung function and circulation. Blood tests and lung function studied also in outpatient control about 1 week after surgery.

The two groups of patients (for respectively normal respiratory therapy and suspected lung protective) compared subsequent terms. Impact on lung function, renal function and circulation as well as the number and severity of any complications compared to assess whether the suspected lung protective ventilator therapy is safe and provides adequate beneficial effect to introduce as standard in the future.

Tissue sampling used in the form of blood tests or urine tests MHP research biobank in the experiment. This tissue will be used for analyzes in the specific project and the tissue will be destroyed after current guidelines for project completion.

Side effects and risks:

There are at every blood sampling a small risk of infection and bleeding. Using standard sterile technique. Blood volume removed by blood tests is max of 250 ml in total. Removing this amount of blood does not entail health risks in patients. There may be discomfort around the injection site, the needle drop is wrong in the arm, but using standard sterile technique and dropped down by experienced personnel. Blood samples for the experiment performed during routine blood sampling equipment as specified in the department's instructions.

For lung studies will in some cases could be detected a certain constriction of the small branches of the airways (bronchi). To determine whether this is a condition may require treatment given ally a spray to suck, which aims to expand the branches in order to improve lung function. This medication can cause slight transient dizziness and palpitations.

Disadvantages:

The additional lung examinations in the study will attempt established in connection with the patient's usual attendance and stay at the hospital to avoid extra visits. There must be calculated some extra time spent for outpatient visits in connection with participation in the trial. There is no economic disadvantages associated with the trial for the patient.

Economic conditions:

There is no economic disadvantages associated with the trial for the patient. Funding for the project will be done through a joint financing by the Urology Department D, Department of Anesthesiology and University Clinic for Kidney disease and high blood pressure, Hospital West and Aarhus University. Research funds will be sought from public and private funds.

Publication of trial results:

The results, both positive and negative findings, will be made published in internationally recognized scientific journal anonymously with no personally identifiable data.

Research Ethics statement:

The project reported to the Ethical Science Council at the Central Denmark Region. Database for the project must be approved by the Data Protection Agency by Region of Central. The project is started only after the approval of these two bodies. The project will comply with applicable GCP rules.

Recruitment of participants:

First contacting the patient about the project via the operator, Urology Department, at the information interview on operation. If the patient wants to get further information about the project handed out written information and project manager contacted.

The written information consists of: Participant Information, consent form, "Information for subjects" and "Your Rights as a test subject in a biomedical research." The patient is informed both in writing and orally on the right and the opportunity to bring legal counsel to informed consent.

The project manager or his representative hold subsequent information interview about 7 days before surgery. This will last approximately 30 minutes. Information being conducted in consultation room at the clinic, where there is no other activity in the allocated room during the interview.

The anesthesia controller or his deputy hold right now usual anesthesia monitoring and ensuring written consent.

At the oral information, patients will be informed that there is a request to participate in a biomedical research. Patients are informed acc. the guidelines in "Guidelines for review, etc. of a biomedical research for the ethics committee system "from the Central Scientific Ethical Committee. Information is provided for the experiment, as listed in Annex 1 "Information for volunteers." The subjects, who wish to participate are advised that, if they wish, can get consideration before submitting their written consent to participate in research is voluntary, and that they will always be able to draw a committed participation back .

The subjects were informed that they will receive information on the results achieved by research reporting on the project if they are interested in this.

Written informed consent given to the project manager or the anesthetic consultant or his deputy in the project in connection with the information interview, journal recording and anesthesia monitoring. The subjects signed concent- and proxy statement, which is kept by the Data Protection Agency guidelines. A copy provided to the subject.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Men
* Indication for robot-assisted radical prostatectomy acc. the department's instructions

Exclusion Criteria:

* Lack of desire to participate
* EGFR <15 ml / min
* BMI> 35 kg / m2
* Former lung surgery
* Known requiring treatment lung disease
* Known heart disease svt NYHA Class III or higher
* Recent AMI within 12 months
* Known neuromuscular disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
PaO2 2 hours postoperatively after 10 minutes of spontaneous respiration of atmospheric air | 10 minutes

SECONDARY OUTCOMES:
Difference in cytokines released from lung tissue measured by IL-6. | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospitalsenheden Vest, Holstebro, Denmark

REFERENCES:
- [Derived] Hoyer S, Mose FH, Ekelof P, Jensen JB, Bech JN. Hemodynamic, renal and hormonal effects of lung protective ventilation during robot-assisted radical prostatectomy, analysis of secondary outcomes from a randomized controlled trial. BMC Anesthesiol. 2021 Aug 5;21(1):200. doi: 10.1186/s12871-021-01401-x. PMID 34348666